CLINICAL TRIAL: NCT07393386
Title: Intrapleural Bupivacaine Analgesia for Postoperative Pain Management After Minimally Invasive Video-Assisted Thoracoscopic Surgery: A Randomized Controlled Trial
Acronym: IBVATS
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Wei Wu, Attending Physician, Department of Anesthesiology, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IDLJ-20251125
Record Dates: First submitted 2026-02-01; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Pain Management
Keywords: Postoperative pain; Thoracoscopic surgery; Intrapleural analgesia
MeSH Terms: conditions — Agnosia; Pain, Postoperative | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 0.25% Bupivacaine Intrapleural Analgesia (Experimental): Participants receive programmed intermittent intrapleural administration of 0.25% bupivacaine via a chest drainage tube connected to a programmed infusion pump for postoperative analgesia following video-assisted thoracoscopic surgery. All participants also receive standard multimodal analgesia, including intravenous patient-controlled analgesia, regional nerve block, and rescue analgesic medications as clinically indicated.
  Interventions: Drug: Bupivacaine 0.25%; Other: Multimodal Analgesia
- 0.125% Bupivacaine Intrapleural Analgesia (Experimental): Participants receive programmed intermittent intrapleural administration of 0.125% bupivacaine via a chest drainage tube connected to a programmed infusion pump for postoperative analgesia following video-assisted thoracoscopic surgery. All participants also receive standard multimodal analgesia, including intravenous patient-controlled analgesia, regional nerve block, and rescue analgesic medications as clinically indicated.
  Interventions: Drug: Bupivacaine 0.125%; Other: Multimodal Analgesia
- Placebo Intrapleural Analgesia (Normal Saline) (Placebo Comparator): Participants receive programmed intermittent intrapleural administration of normal saline via a chest drainage tube connected to a programmed infusion pump as a placebo control for postoperative analgesia following video-assisted thoracoscopic surgery. All participants also receive standard multimodal analgesia, including intravenous patient-controlled analgesia, regional nerve block, and rescue analgesic medications as clinically indicated.
  Interventions: Drug: Normal Saline; Other: Multimodal Analgesia

INTERVENTIONS:
Drug: Bupivacaine 0.125% — Bupivacaine 0.125% is administered intrapleurally via a chest drainage tube connected to a programmed infusion pump, using a programmed intermittent dosing regimen for postoperative analgesia following video-assisted thoracoscopic surgery.
  Arms: 0.125% Bupivacaine Intrapleural Analgesia
Drug: Bupivacaine 0.25% — Bupivacaine 0.25% is administered intrapleurally via a chest drainage tube connected to a programmed infusion pump, using a programmed intermittent dosing regimen for postoperative analgesia following video-assisted thoracoscopic surgery.
  Arms: 0.25% Bupivacaine Intrapleural Analgesia
Drug: Normal Saline — Normal saline is administered intrapleurally via a chest drainage tube connected to a programmed infusion pump, using a programmed intermittent dosing regimen as a placebo control for postoperative analgesia following video-assisted thoracoscopic surgery.
  Arms: Placebo Intrapleural Analgesia (Normal Saline)
Other: Multimodal Analgesia — All participants receive standard multimodal analgesia, including intravenous patient-controlled analgesia, regional nerve block, and rescue analgesic medications as clinically indicated, in addition to the assigned intrapleural intervention.

SUMMARY:
Postoperative pain is common after video-assisted thoracoscopic surgery (VATS), with pleural irritation caused by chest tube placement being a major contributor. Inadequate pain control may impair respiratory function, delay postoperative recovery, and increase the risk of complications. However, effective and targeted analgesic strategies specifically addressing chest tube-related pain remain limited.

This is a single-center, prospective, randomized, double-blind, placebo-controlled superiority trial designed to evaluate the efficacy and safety of programmed intermittent intrapleural administration of bupivacaine at different concentrations for postoperative analgesia after VATS. A total of 249 patients undergoing VATS will be randomly assigned in a 1:1:1 ratio to receive intrapleural injections of 0.25% bupivacaine, 0.125% bupivacaine, or normal saline. The primary outcome is pain intensity during coughing within 48 hours after surgery. Secondary outcomes include pain intensity at rest, plasma bupivacaine concentrations, quality of postoperative recovery, cumulative opioid consumption, and postoperative inflammatory marker levels.

This study aims to provide evidence to inform analgesic strategies for chest tube-related pain following VATS and to clarify the optimal use and safety profile of intrapleural bupivacaine.

DETAILED DESCRIPTION:
Postoperative pain is common after video-assisted thoracoscopic surgery (VATS), with pleural irritation caused by chest tube placement being a major contributor. Inadequate pain control may impair respiratory function, delay postoperative recovery, and increase the risk of complications. However, effective and targeted analgesic strategies specifically addressing chest tube-related pain remain limited.

This is a single-center, prospective, randomized, double-blind, placebo-controlled superiority trial designed to evaluate the efficacy and safety of programmed intermittent intrapleural administration of bupivacaine at different concentrations for postoperative analgesia after VATS. A total of 249 patients undergoing VATS will be randomly assigned in a 1:1:1 ratio to receive intrapleural injections of 0.25% bupivacaine, 0.125% bupivacaine, or normal saline. The primary outcome is pain intensity during coughing within 48 hours after surgery. Secondary outcomes include pain intensity at rest, plasma bupivacaine concentrations, quality of postoperative recovery, cumulative opioid consumption, and postoperative inflammatory marker levels.

This study aims to provide evidence to inform analgesic strategies for chest tube-related pain following VATS and to clarify the optimal use and safety profile of intrapleural bupivacaine.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for elective video-assisted thoracoscopic surgery
2. Age≥18 years
3. American Society of Anesthesiologists (ASA) physical status classification I-III

Exclusion Criteria:

1. Pregnancy or breastfeeding
2. History of chronic pain
3. History of alcohol or opioid dependence
4. Significant cardiopulmonary dysfunction, including heart failure or severe cardiac conduction abnormalities
5. Coexisting central nervous system disorders
6. Hepatic or renal dysfunction
7. Known hypersensitivity to local anesthetics or opioids
8. Local infection at or near the planned site of regional anesthesia, or systemic infection
9. Language impairment or difficulty in communication
10. Refusal to participate in the study or refusal to use patient-controlled analgesia
11. Concurrent participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Area Under the Curve of Pain Intensity During Coughing | 1, 2, 6, 12, 24, 36, and 48 hours postoperatively
  Pain intensity during coughing will be assessed using the Numerical Rating Scale (NRS; range 0-10). The area under the curve (AUC) of NRS pain scores will be calculated based on repeated measurements to reflect overall pain burden during the first 48 hours after surgery. Pain assessments will be performed by trained study evaluators.

SECONDARY OUTCOMES:
Area Under the Curve of Resting Pain Intensity | 1, 2, 6, 12, 24, 36, and 48 hours postoperatively
  Pain intensity at rest will be assessed using the Numerical Rating Scale (NRS; range 0-10). The area under the curve (AUC) of NRS pain scores will be calculated based on repeated assessments to evaluate cumulative resting pain during the first 48 hours after surgery. Assessments will be performed by trained study evaluators.
Postoperative Opioid Consumption | Up to 48 hours postoperatively
  Total opioid consumption within the first 48 hours after surgery will be recorded and analyzed.
Quality of Recovery | Baseline (preoperative), 24 hours, and 48 hours postoperatively
  Postoperative recovery quality will be assessed using the 40-item Quality of Recovery questionnaire (QoR-40), which evaluates multiple domains of postoperative recovery.

OTHER OUTCOMES:
Plasma Bupivacaine Concentration | From pre-administration to 48 hours postoperatively
  Plasma concentrations of bupivacaine will be measured to assess systemic exposure following intrapleural administration. Venous blood samples will be collected at predefined time points and analyzed using validated analytical methods. Concentration-time data will be used to characterize the pharmacokinetic profile.
Patient Satisfaction With Pain Management | 48 hours postoperatively
  Patient satisfaction with postoperative pain management will be assessed using a 5-point Likert scale ranging from 1 (very dissatisfied) to 5 (very satisfied), reflecting overall satisfaction with pain control.
Rescue Analgesic Consumption | Up to 48 hours postoperatively
  Total consumption of rescue analgesic medications administered within the first 48 hours after surgery will be recorded and analyzed.
Postoperative Systemic Inflammatory Response | Baseline (preoperative) and 24 hours postoperatively
  The postoperative systemic inflammatory response will be assessed as a composite evaluation based on venous blood samples. This assessment will characterize the overall inflammatory response by integrating multiple inflammatory components, including serum cytokine levels (IL-6, IL-8, IL-12, TNF-α), C-reactive protein (CRP), and cellular inflammation indices derived from complete blood count data, including the systemic immune-inflammation index (SII), neutrophil-to-lymphocyte ratio (NLR), and platelet-to-lymphocyte ratio (PLR).
Adverse Events | From informed consent to hospital discharge (serious adverse events followed up to 30 days post-discharge)
  All adverse events will be recorded from the time of informed consent through hospital discharge. Adverse event severity will be graded according to the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0, and events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA), version 26.1. Serious adverse events will be followed until resolution, stabilization, or up to 30 days after hospital discharge, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
De identified individual participant data and related study documents (e.g., study protocol, statistical analysis plan) will be made available upon reasonable request after the completion of the study. Researchers interested in data access may submit a proposal to the principal investigator via email. The proposal should include a detailed research plan and data analysis proposal. Data will be provided following review and approval by the study team. Contact Email: 18621710790@163.com
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Supporting documentation will be made available beginning 12 months after publication of the primary study results and will remain available for 5 years thereafter.
Access Criteria: De-identified individual participant data that underlie the results reported in the primary publication, as well as the study protocol and statistical analysis plan, will be available to qualified researchers. Requests must be submitted to the principal investigator and will be reviewed on a case-by-case basis. Access will be granted for scientifically sound proposals and subject to approval by the study team and the execution of a data use agreement.